CLINICAL TRIAL: NCT00687310
Title: Does Tailored Education in Asthma Care Help Improve Patient Satisfaction, Adherence, and Quality of Life (TEACH) Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Gloria Jordana - Scientific Director-GI/RITA, AstraZeneca Canada Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D5890L00018
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma education; satisfaction adherence; Quality of Life; PIKO meter cluster; Symbicort® Turbuhaler®
MeSH Terms: conditions — Asthma | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Educational Intervention At the initial visit (Visit 1), patients in the educational intervention group will complete a short Needs Assessment Questionnaire to help the investigator/nurse determine which section(s) of the tailored patient education booklet to give to, educate, and provide instruction on to the patient. This may, at the discretion of the investigator, include providing their patient with a peak flow meter and instructions on its use.Visit 2 will be scheduled for 1-month after the Visit 1 for the education intervention group. All educational materials provided at Visit 1 will be reviewed with the patient at Visit 2. The investigator/nurse will reassess the patient's use of the Turbuhaler® and asthma treatment plan. Patients will also be asked about any adverse events that may have occurred since Visit 1 and/or are observed at Visit 2. Once Visit 2 is completed with the patient, the investigator/nurse will complete the Educator Satisfaction Questionnaire.
  Interventions: Behavioral: Educational intervention

INTERVENTIONS:
Behavioral: Educational intervention — Tailored asthma education based on needs assessment

SUMMARY:
The primary purpose of this study is to assess whether tailored patient education for patients on Symbicort® Turbuhaler® therapy improves patient satisfaction, adherence and Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of asthma.
* Patients with asthma, where the use of Symbicort® Turbuhaler® is indicated and would have been prescribed by the investigator as part of usual care.
* Patient who have public or private insurance coverage for Symbicort® Turbuhaler® or are willing to pay for this medication for the duration of the trial.

Exclusion Criteria:

* Patients who have been treated wth Symbicort® Turbuhaler® in the preceding 3 months.
* A history of smoking [i.e., 10 pack-years where one pack-year equals one pack (20 cigarettes) per day for one year, or equivalent].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2005-12; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Patient's satisfaction with asthma education | At the initial visit (Visit 1) and during the final call (Call 2) or at the time of premature discontinuation from the trial.

SECONDARY OUTCOMES:
Mini-asthma Quality of Life questionnaire | Visit 1 and during calls 1 and 2
Asthma control parameters | At baseline, as well as during Call 1 and Call 2 for both the usual care group and the enducational intervention group.
PIKO meter usage assessment | During the Call 2 to the educational intervention group subjects who received the PIKO meter during their educational session.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McIvor, M.D., M.Sc., FRCP(E), FRCP(C), Principal Investigator — McMaster University; Christopher Licskai, M.D., FRCPC, Principal Investigator — University of Ontario London Ontario Canada; Alan Kaplan, M.D., CCFP, CCFP(E.M.), Principal Investigator — York Central Hospital, Richmond Hill, Ontario Canada